CLINICAL TRIAL: NCT02721862
Title: Effectiveness of Ursodeoxycholic Acid Use in the Prevention of Gallstone Formation After Sleeve Gastrectomy: A Prospective Randomized Multicenter Placebo-Controlled Trial
Brief Title: Effectiveness of Ursodeoxycholic Acid Use in the Prevention of Gallstone Formation After Sleeve Gastrectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ramzi Alami, MD, FACS, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SUR.RA.01
Record Dates: First submitted 2016-03-18; First posted 2016-03-29 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2016-03

CONDITIONS: Cholelithiasis
Keywords: gallstones; cholelithiasis; sleeve gastrectomy
MeSH Terms: conditions — Cholelithiasis; Gallstones | interventions — Ursodeoxycholic Acid; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): This arm will include 50 patients who, at baseline ultrasound, have no gallbladder pathology and have no previous cholecystectomy. Those patients will be taking an oral drug (Ursodeoxycholic Acid 250mg) twice daily for a period of six months and undergoing a total of three gallbladder ultrasounds (at 6 months, at 12 months, and at 18 months) to check for gallstones.
  Interventions: Drug: Ursodeoxycholic Acid; Radiation: Gallbladder Ultrasound
- Control (Placebo Comparator): This arm will include 50 patients who, at baseline ultrasound, have no gallbladder pathology and have no previous cholecystectomy. Those patients will be taking a placebo, that is dispensed from the pharmacy and having the same color as the ursodeoxycholic acid 250mg, twice daily for a period of six months and undergoing a total of three gallbladder ultrasounds (at 6 months, at 12 months, and at 18 months) to check for gallstones.
  Interventions: Drug: Placebo; Radiation: Gallbladder Ultrasound

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Ursodeoxycholic acid, is FDA approved for the reduction in gallstone formation in obese patients undergoing rapid weight loss.Ursofalk is indicated in the treatment of primary biliary cirrhosis (PBC) and for the dissolution of radiolucent gallstones in patients with a functioning gall bladder.
  Other Names: Ursofalk
  Arms: Experimental
Drug: Placebo — The placebo has the same color and size as the ursodeoxycholic acid 250 mg pill
  Other Names: Sugar pill
  Arms: Control
Radiation: Gallbladder Ultrasound — Each patient will undergo a total of three abdominal ultrasounds (at 6 months, at 12 months, and at 18 months after sleeve gastrectomy) to check for gallstones. Patients should be gallstone free on an initial ultrasound to satisfy the study inclusion criteria. Ultrasound testing is radiation free and does not pose any additional risk to the subjects.

SUMMARY:
This is a randomized double-blind placebo-controlled trial with a total of 100 patients who are free of gallstones at baseline. The study involves taking an oral drug (Ursodeoxycholic Acid 250mg) or a placebo twice daily for a period of six months and undergoing a total of three abdominal ultrasounds (at 6 months, at 12 months, and at 18 months) to check for gallstones.

DETAILED DESCRIPTION:
A significant proportion of patients are known to develop gallstones during the phase of rapid weight loss after bariatric surgery. A small percentage of these patients develop symptoms such as abdominal pain, nausea, vomiting, and occasionally more serious symptoms relating to gallbladder disease. Those patients may require surgery for the removal of their gallbladder even though the risks of gallbladder surgery are increased in this patient group.

The investigators would like to provide patients who have undergone Laparoscopic Sleeve Gastrectomy a drug that will reduce the risk of developing gallstones during the phase of rapid weight loss after surgery. The drug, Ursodeoxycholic acid, is FDA approved for the reduction in gallstone formation in obese patients undergoing rapid weight loss but has never been proven effective, by randomized controlled studies, in the subgroup of obese patients undergoing Laparoscopic Sleeve Gastrectomy. If proven so, the investigators intend to influence the current practice such that all patients are offered Ursodeoxycholic Acid for the reduction of gallstone formation and their complications following Laparoscopic Sleeve Gastrectomy.

In this randomized double-blind placebo-controlled trial, the subjects will be approached by the principal investigator in the clinic with information about taking part in this study, after the decision is made to undergo Laparoscopic Sleeve Gastrectomy for weight loss. The surgeon will answer any questions then and thereafter. The investigators will clarify that participation is voluntary and will not alter routine care whether the patient participates or not. The study involves taking an oral drug (Ursodeoxycholic Acid 250mg) twice daily for a period of six months and undergoing a total of three abdominal ultrasounds (at 6 months, at 12 months, and at 18 months) to check for gallstones. Patients should be gallstone free on an initial ultrasound to satisfy the study inclusion criteria. Ultrasound testing is radiation free and does not pose any additional risk to the subjects.

A total of 100 patients need to be recruited. The sample is comparable to current studies and is sufficient to prove or disprove the hypothesis with low risk of error (ref). The patients will either receive placebo or the drug under study, the placebo being dispensed from the pharmacy and having the same color as the ursodeoxycholic acid. The principal investigator and the radiologists measuring the result will be blinded to whether the subject receives the drug or placebo.

The study needs to involve human subjects so that the results will be applicable to human subjects. The risk is small because the drug is FDA approved with 13 years post-marketing experience for related indications and is known to be well tolerated. All efforts will be made to protect the privacy and confidentiality of the subjects including protecting their personal information by removing identifiers from data records and storing the identifying codes in a separate location, with all study material under password protection or lock and key at all times.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (body mass index > 35 kg/m2) undergoing laparoscopic sleeve gastrectomy as a primary treatment for their obesity.
* No gallstone disease on initial ultrasounds
* No previous cholecystectomy

Exclusion Criteria:

* Bariatric patients with gallbladder stones on baseline ultrasound examination.
* Patients with a previous cholecystectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-09 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of gallstone formation after laparoscopic sleeve gastrectomy | At 6 months to 18 months after laparoscopic sleeve gastrectomy
  Patients in both arms will undergo a total of three abdominal ultrasounds after their bariatric surgery (at 6 months, at 12 months, and at 18 months) to check for gallstones. Once gallstone formation is detected at any of these time points, no additional ultrasounds will be done and the incidence of gallstone formation (Percentage of patients with gallstone formation on ultrasound) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi S. Alami, Md, FACS, Principal Investigator — American University of Beirut Medical Center
Locations (2):
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut
  - Makassed General Hospital, Beirut

IPD SHARING:
Plan to Share IPD: Undecided